CLINICAL TRIAL: NCT03757286
Title: Aesthetic Reconstruction of Onco-surgical Maxillary Defects Using Free Scapular Flap With and Without CAD/CAM Customized Osteotomy Guide (A Randomized Controlled Clinical Trial)
Brief Title: Aesthetic Reconstruction of Onco-surgical Maxillary Defects Using FSF With and Without CAD/CAM Customized Cutting Guide
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Salah Mohammed Al-Wadeai, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 654
Record Dates: First submitted 2018-11-27; First posted 2018-11-28 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Maxillary Tumors
Keywords: maxillary tumors resection\ reconstruction; CAD\CAM; osteotomy, cutting guide; aesthetic; operation time; free scapular flap

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Because the two interventions used in this trial are easily recognized by the participants and the investigator, neither the investigator nor the participant can be blinded. But, assessor and the statistician will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSF with CAD\CAM customized cutting guide (Experimental): Maxillary reconstruction using free scapular flap with CAD/CAM customized osteotomy guide.
  Interventions: Procedure: FSF with CAD\CAM customized cutting guide
- FSF without customized cutting guide (Active Comparator): maxillary reconstruction using free scapular flap without customized osteotomy guide. CAD/CAM 3D model for maxilla will be used.
  Interventions: Procedure: FSF without customized cutting guide

INTERVENTIONS:
Procedure: FSF with CAD\CAM customized cutting guide — This began with the acquisition of a high-resolution CT scan of the patient's maxilla and scapula. The CT scan will be sent to the modeling company that produce 3D autoclavable models and cutting guides to be used during resection and scapular harvesting as well as a model of the final reconstructed maxilla.
  surgery will performed by two surgical teams one for tumor resection and the other harvesting the flap.
  access to the maxilla was obtained and the cutting guides were secured in the planned position; the cuts were completed. The scapular guides were secured to the harvested scapula to replicate the cuts that were planned previously.
  The scapula and plate will be fixed and pedicle anastomosis is performed. the operation then completed with soft tissue reconstruction.
  Arms: FSF with CAD\CAM customized cutting guide
Procedure: FSF without customized cutting guide — This began with the acquisition of a high-resolution CT scan of the patient's maxilla .
  The C.T scan will be sent to the modeling company for planning three-dimensional model of the maxilla. autoclavable model will be prepared to be used during the workflow for plate reshaping to conforme the prices position of the maxilla.
  surgery will performed in a single step by two surgical teams, one for cervicofacial resection and the other for harvesting the flap.
  Resection-reconstruction then performed in aconventional surgical manner with microvascular anastomosis. finally the operation will be completed with soft tissue reconstruction as needed.
  Arms: FSF without customized cutting guide

SUMMARY:
The aim of the study is to compare aesthetic results and operation time of Free Scapular flap with and without CAD/CAM customized osteotomy guide for reconstruction of maxillary Defects.

DETAILED DESCRIPTION:
Maxillofacial defects create unique challenges for the reconstructive surgeon, often involving bony and soft tissue components of the midface. Surgical reconstruction following maxillectomy is currently a topic of interest for reconstructive head and neck surgeons. maxillary defects were reconstructed with maxillofacial prosthetics including obturation. While the latter is an effective reconstruction. Over the past two decades, there has been increasing interest in the use of free tissue transfers of bone to reconstruct the maxilla.

Scapular flap It is an excellent candidate for maxillectomy defects because of its unique feature, which is characterized by additional skin paddles or muscles. and can be harvested along with a part of the scapular bone for bony reconstruction

Traditional reconstructive techniques often lead to suboptimal reconstructions due to inexact planning, poor communication between the resective and reconstructive teams or surgical difficulties in adjusting a free flap and osteosynthesis plates into a three-dimensional (3D) defect without the help of any templates or surgical guides The advent of 3D modeling in head and neck reconstruction has allowed surgeons to improve upon functional and aesthetic outcomes, which are crucial to patient satisfaction and can be difficult to achieve in maxillectomy defects The cutting guides used or not used, however debate still present for its benefits and worth for patient and surgeon. current study to evaluate how such virtual planning with using of customized cutting guide is effective and worth for patient aesthetic and operation time.

our priori-hypothesis is that utilization CAD/CAM assisted with customized osteotomy guide is not related to an altered result regarding aesthetic outcome and operation time in patient undergoing maxillary reconstruction using free scapular flap.

In order to test this hypothesis, we will compare aesthetic outcome and operation time in group of patients receive FSF by CAD/CAM-assisted with customized osteotomy guide to results of another group of patients receive FSF but without customized osteotomy guide. only model will be performed as conventional method aiding in reshaping of reconstruction plate which is another well-established concept of management of maxillary defect.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by tumor involving Maxillary bone.

Exclusion Criteria:

* Patients having poor oncological prognosis
* Patients with poor performance status together with other relative or absolute vascular contraindication.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Aesthetic | at least three months postoperative
  aesthetic outcome will be measured objectively by computerized digital analysis as differential angle and differential area of reconstructed to other side of maxilla.subjectively will be evaluated using VAS.

SECONDARY OUTCOMES:
operation time | intraoperative
  operation time will be recorded intraoperatively in the surgery day as total operation time and ischemic time.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Al-wadeai, Phd. student, Principal Investigator — Cairo University
Locations (1):
- Faculity of Dentistry-Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Alwadeai MS, Al-Aroomy LA, Shindy MI, Amin AA, Zedan MH. Aesthetic reconstruction of onco-surgical maxillary defects using free scapular flap with and without CAD/CAM customized osteotomy guide. BMC Surg. 2022 Oct 19;22(1):362. doi: 10.1186/s12893-022-01811-9. PMID 36261822